CLINICAL TRIAL: NCT02348918
Title: A Phase 2 Randomized, Controlled, Double-Masked, Multicenter Clinical Trial Designed to Evaluate the Safety and Exploratory Efficacy of Luminate® (ALG-1001) as Compared to Avastin® in the Treatment of Diabetic Macular Edema (DME)
Brief Title: Phase 2 Randomized Clinical Trial of Luminate® as Compared to Avastin® in the Treatment of Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allegro Ophthalmics, LLC (Industry)
Collaborators: Trial Runners, LLC (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DME 202B
Record Dates: First submitted 2015-01-12; First posted 2015-01-28 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — risuteganib; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Luminate 1.0mg group (Active Comparator): Stage 1- Luminate 1.0 mg intravitreal injection administered at baseline (Day 0), 4 weeks and 8 weeks with prn Luminate injection at week 20 for a total of at least 3 and no more than 4 Luminate injections. Sham injections will be performed at weeks 12 and 16 and may also be performed at week 20 if prn Luminate is not required; sham laser treatment will be administered at baseline and at 16 weeks.
  Interventions: Drug: Luminate 1.0mg
- Luminate 2.0mg group (Active Comparator): Stage 1 -Luminate 2.0 mg intravitreal injection administered at baseline (Day 0), 4 weeks and 8 weeks with prn Luminate injection at week 20 for a total of at least 3 and no more than 4 Luminate injections. Sham injections will be performed at weeks 12 and 16 and may also be performed at week 20 if prn Luminate is not required; sham laser treatment will be administered at baseline and at 16 weeks.
  Interventions: Drug: Luminate 2.0mg
- Luminate 3.0mg group (Active Comparator): Stage 1- Luminate 3.0 mg intravitreal injection administered at baseline (Day 0), 4 weeks and 8 weeks with prn Luminate injection at week20 for a total of at least 3 and no more than 4 Luminate injections. Sham injections will be performed at weeks 12 and 16 and may also be performed at week 20 if prn Luminate is not required; sham laser treatment will be administered at baseline and at 16 weeks.
  Interventions: Drug: Luminate 3.0mg
- Avastin® group (Active Comparator): Stage 1- Avastin 1.25 mg intravitreal injection administered at baseline (Day 0), 4 weeks and 8 weeks with prn Avastin injection at weeks 12, 16, or 20 for a total of at least 3 and up to 6 Avastin injections. Sham injections may be performed at weeks 12, 16, and 20 if prn Avastin is not required.
  Interventions: Drug: Avastin
- Avastin then Luminate 1.0 mg IVT + sham injection (Active Comparator): Stage 2 - Week 0 (Baseline): Avastin 1.25 mg IVT Weeks 1, 4 and 8: Luminate 1.0 mg IVT + sham injection Weeks 12 and 16: Sham IVT
  Interventions: Drug: Luminate 1.0mg; Drug: Avastin
- Avastin then Luminate 0.5 mg IVT + sham injection (Active Comparator): Stage 2- Week 0 (Baseline); Avastin 1.25 mg IVT Weeks 1, 4 and 8: Luminate 0.5 mg IVT + sham injection Weeks 12 and 16: Sham IVT
  Interventions: Drug: Avastin; Drug: Luminate 0.5mg
- Sham then Luminate 1.0 mg + Avastin 1.25 mg IVT (Active Comparator): Stage 2 : Week 0 (Baseline): Sham IVT Weeks 1, 4 and 8: Luminate 1.0 mg + Avastin 1.25 mg IVT Weeks 12 and 16: Sham IVT
  Interventions: Drug: Luminate 1.0mg; Drug: Avastin
- Sham then Luminate 0.5 mg IVT + Avastin 1.25 mg IVT (Active Comparator): Stage 2 : Week 0: Sham IVT Weeks 1, 4 and 8: Luminate 0.5 mg IVT + Avastin 1.25 mg IVT Weeks 12 and 16: Sham IVT
  Interventions: Drug: Avastin; Drug: Luminate 0.5mg
- Avastin 1.25 mg + Sham IVT (Active Comparator): Stage 2 : Week 0 (Baseline): Sham IVT Weeks 1, 4 and 8: Avastin 1.25 mg + Sham IVT Weeks 12 and 16: Avastin PRN
  Interventions: Drug: Luminate 0.5mg

INTERVENTIONS:
Drug: Luminate 1.0mg
  Other Names: ALG-1001
  Arms: Avastin then Luminate 1.0 mg IVT + sham injection; Luminate 1.0mg group; Sham then Luminate 1.0 mg + Avastin 1.25 mg IVT
Drug: Luminate 2.0mg
  Other Names: ALG-1001
  Arms: Luminate 2.0mg group
Drug: Luminate 3.0mg
  Other Names: ALG-1001
  Arms: Luminate 3.0mg group
Drug: Avastin
  Other Names: bevacizumab
  Arms: Avastin then Luminate 0.5 mg IVT + sham injection; Avastin then Luminate 1.0 mg IVT + sham injection; Avastin® group; Sham then Luminate 0.5 mg IVT + Avastin 1.25 mg IVT; Sham then Luminate 1.0 mg + Avastin 1.25 mg IVT
Drug: Luminate 0.5mg
  Other Names: ALG-1001
  Arms: Avastin 1.25 mg + Sham IVT; Avastin then Luminate 0.5 mg IVT + sham injection; Sham then Luminate 0.5 mg IVT + Avastin 1.25 mg IVT

SUMMARY:
A Phase 2 Multi center, Randomized, Controlled, Double-Masked Clinical Trial Designed To Evaluate The Safety And Exploratory Efficacy Of Luminate® (Alg-1001) As Compared To Avastin® In The Treatment Of Diabetic Macular Edema

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of Luminate® (ALG-1001) as compared to Avastin® in patients with diabetic macular edema

- Stage 1: 120 eligible subjects with DME will be enrolled and randomized to one of 4 treatment groups at an allocation ratio of 1:1:1:1, i.e., one of three doses (1.0 mg, 2.0 mg and 3.0 mg) of Luminate intravitreal injection or Avastin intravitreal injection. Subjects will be followed monthly for 24 weeks (6 months).

Stage 2 (select sites): 75 eligible subjects with DME will be enrolled and randomized to one of 5 treatment groups at an allocation ratio of 1:1:1:1:1; i.e., one of 2 doses of Luminate intravitreal injection or Avastin intravitreal injection (0.5 mg and 1.0 mg). Subjects will be followed monthly for 20 weeks (5 months).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older.
* Study eye with clinically significant diabetic macular edema (DME) with central subfield thickness ≥ 350µm on spectral domain OCT
* Best corrected visual acuity (BCVA) of 20/50 to 20/320 ETDRS equivalent (65 letters to 23 letters) in the study eye, with BCVA decrement primarily attributable to DME.
* Treatment naïve, i.e., no previous anti-VEGF treatment in the study eye or no anti-VEGF treatment in the 45 days prior to study enrollment.
* In the investigator's opinion, the subject still has significant intraretinal fluid with room for improvement in both macular edema and BCVA.
* Intra-Ocular Pressure (IOP) is under control (i.e., IOP

  ≤ 25 mm in the study eye) and study eye is not receiving any IOP lowering drops.
* Willing and able to return for all study visits.
* Able to meet the extensive post-op evaluation regimen.
* Understands and signs the informed consent form.

Exclusion Criteria:

* Active proliferative diabetic retinopathy (PDR) in the study eye such as NVE, NVD, vitreous hemorrhage, or neovascular glaucoma.
* Uncontrolled hypertension defined as systolic >180 mmHg or > 160 mmHg on 2 consecutive measurements or diastolic > 100 mmHg on optimal medical regimen
* Screening HgA1c blood test > 10.0
* Focal laser photocoagulation or intravitreal/periocular steroids of any type in the study eye within the last 90 days prior to study enrollment.
* A history of intravitreal anti-VEGF injection of any type in the study eye within the last 45 days prior to study enrollment.
* History of rhegmatogenous retinal detachment, retinal tear(s), or traction retinal detachments in the study eye.
* Epiretinal membrane and/or vitreomacular traction in the study eye as determined by the central reading center.
* Previous pars plana vitrectomy in the study eye
* Any intraocular surgery in the study eye within the last 90 days prior to study enrollment.
* YAG laser treatment in the study eye in last 30 days prior to study enrollment.
* High myopia in the study eye, with a spherical equivalent of >8.00D at screening
* Other ocular pathologies that in the investigator's opinion would interfere with the subject's vision in the study eye.
* Chronic or recurrent uveitis.
* Ongoing ocular infection or inflammation in either eye.
* A history of cataract surgery complications/vitreous loss in the study eye.
* Congenital eye malformations in the study eye.
* A history of penetrating ocular trauma in the study eye.
* Mentally handicapped.
* Pregnant female, as determined for women less than 60 years old by a positive urine pregnancy test during the screening window.
* Nursing female.
* Currently participating in any other clinical research study.
* Contraindication to the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicken Karageozian, Study Director — Cheif Medical Officer
Locations (17):
- United States (17):
  - Associated Retina Consultants, Phoenix, Arizona
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - West Coast Retina, San Francisco, California
  - Orange County Retina Medical Group, Santa Ana, California
  - New England Retina Associates, New London, Connecticut
  - Florida Eye Clinic, Altamonte Springs, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Wilmer Eye Institute at John Hopkins University, Baltimore, Maryland
  - TLC Eye Group, Jackson, Michigan
  - Island Retina, Shirley, New York
  - Charlotte EENT Associates, Charlotte, North Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Austin Retina Associates, Austin, Texas
  - Retina Consultant of Houston, Houston, Texas
  - Spokane Eye Clinical Research, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Luminate 1.0mg Group: Stage 1- Luminate 1.0 mg intravitreal injection administered at baseline (Day 0), 4 weeks and 8 weeks with prn Luminate injection at week 20 for a total of at least 3 and no more than 4 Luminate injections. Sham injections will be performed at weeks 12 and 16 and may also be performed at week 20 if prn Luminate is not required; sham laser treatment will be administered at baseline and at 16 weeks.
  Luminate 1.0mg
- Luminate 2.0mg Group: Stage 1 -Luminate 2.0 mg intravitreal injection administered at baseline (Day 0), 4 weeks and 8 weeks with prn Luminate injection at week 20 for a total of at least 3 and no more than 4 Luminate injections. Sham injections will be performed at weeks 12 and 16 and may also be performed at week 20 if prn Luminate is not required; sham laser treatment will be administered at baseline and at 16 weeks.
  Luminate 2.0mg
- Luminate 3.0mg Group: Stage 1- Luminate 3.0 mg intravitreal injection administered at baseline (Day 0), 4 weeks and 8 weeks with prn Luminate injection at week20 for a total of at least 3 and no more than 4 Luminate injections. Sham injections will be performed at weeks 12 and 16 and may also be performed at week 20 if prn Luminate is not required; sham laser treatment will be administered at baseline and at 16 weeks.
  Luminate 3.0mg
- Avastin® Group: Stage 1- Avastin 1.25 mg intravitreal injection administered at baseline (Day 0), 4 weeks and 8 weeks with prn Avastin injection at weeks 12, 16, or 20 for a total of at least 3 and up to 6 Avastin injections. Sham injections may be performed at weeks 12, 16, and 20 if prn Avastin is not required.
  Avastin
- Avastin Then Luminate 1.0 mg IVT + Sham Injection: Stage 2 - Week 0 (Baseline): Avastin 1.25 mg IVT Weeks 1, 4 and 8: Luminate 1.0 mg IVT + sham injection Weeks 12 and 16: Sham IVT
  Luminate 1.0mg
  Avastin
- Avastin Then Luminate 0.5 mg IVT + Sham Injection: Stage 2- Week 0 (Baseline); Avastin 1.25 mg IVT Weeks 1, 4 and 8: Luminate 0.5 mg IVT + sham injection Weeks 12 and 16: Sham IVT
  Avastin
  Luminate 0.5mg
- Sham Then Luminate 1.0 mg + Avastin 1.25 mg IVT: Stage 2 : Week 0 (Baseline): Sham IVT Weeks 1, 4 and 8: Luminate 1.0 mg + Avastin 1.25 mg IVT Weeks 12 and 16: Sham IVT
  Luminate 1.0mg
  Avastin
- Sham Then Luminate 0.5 mg IVT + Avastin 1.25 mg IVT: Stage 2 : Week 0: Sham IVT Weeks 1, 4 and 8: Luminate 0.5 mg IVT + Avastin 1.25 mg IVT Weeks 12 and 16: Sham IVT
  Avastin
  Luminate 0.5mg
- Avastin 1.25 mg + Sham IVT: Stage 2 : Week 0 (Baseline): Sham IVT Weeks 1, 4 and 8: Avastin 1.25 mg + Sham IVT Weeks 12 and 16: Avastin PRN
  Luminate 0.5mg
Period: Overall Study
Arm/Group | Luminate 1.0mg Group | Luminate 2.0mg Group | Luminate 3.0mg Group | Avastin® Group | Avastin Then Luminate 1.0 mg IVT + Sham Injection | Avastin Then Luminate 0.5 mg IVT + Sham Injection | Sham Then Luminate 1.0 mg + Avastin 1.25 mg IVT | Sham Then Luminate 0.5 mg IVT + Avastin 1.25 mg IVT | Avastin 1.25 mg + Sham IVT
Started | 39 | 33 | 42 | 24 | 19 | 17 | 13 | 16 | 15
Completed | 39 | 33 | 42 | 24 | 19 | 17 | 13 | 16 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Luminate 1.0mg Group | Luminate 2.0mg Group | Luminate 3.0mg Group | Avastin® Group | Avastin Then Luminate 1.0 mg IVT + Sham Injection | Avastin Then Luminate 0.5 mg IVT + Sham Injection | Sham Then Luminate 1.0 mg + Avastin 1.25 mg IVT | Sham Then Luminate 0.5 mg IVT + Avastin 1.25 mg IVT | Avastin 1.25 mg + Sham IVT | Total
Number analyzed (Participants) | 39 | 33 | 42 | 24 | 19 | 17 | 13 | 16 | 15 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 29 | 15 | 10 | 10 | 10 | 12 | 9 | 135
  >=65 years | 18 | 14 | 13 | 9 | 9 | 7 | 3 | 4 | 6 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.05) | 61 (9.91) | 63.8 (9.45) | 60.3 (8.83) | 67.1 (10.47) | 65.5 (9.41) | 60.1 (10.92) | 60.5 (8.29) | 62.1 (9.35) | 62.3 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 13 | 17 | 6 | 10 | 12 | 7 | 8 | 10 | 106
  Male | 16 | 20 | 25 | 18 | 9 | 5 | 6 | 8 | 5 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 33 | 29 | 38 | 17 | 17 | 15 | 7 | 13 | 12 | 181
  Black or African American | 4 | 1 | 3 | 3 | 1 | 1 | 5 | 1 | 2 | 21
  Asian | 1 | 1 | 0 | 3 | 0 | 1 | 1 | 2 | 0 | 9
  Other | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 5
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 33 | 42 | 24 | 19 | 17 | 13 | 16 | 15 | 218

OUTCOME MEASURES:

1. Primary Outcome: Change in BCVA at Week 24
Description: Primary efficacy outcome is BCVA changes at Week 24 as compared to baseline
Time Frame: Value of 24 Weeks minus baseline value
Measure: Mean (Standard Error); unit: Letters on ETDRS eye chart
Arm/Group | Luminate 1.0mg Group | Luminate 2.0mg Group | Luminate 3.0mg Group | Avastin® Group | Avastin Then Luminate 1.0 mg IVT + Sham Injection | Avastin Then Luminate 0.5 mg IVT + Sham Injection | Sham Then Luminate 1.0 mg + Avastin 1.25 mg IVT | Sham Then Luminate 0.5 mg IVT + Avastin 1.25 mg IVT | Avastin 1.25 mg + Sham IVT
Number analyzed (Participants) | 39 | 33 | 42 | 24 | 19 | 17 | 13 | 16 | 15
Letters on ETDRS eye chart | 5.2 (3) | 2.7 (3) | -1.5 (3) | 7 (3) | 7.1 (3) | 4.6 (3) | 1.4 (3) | 3.9 (3) | 6.7 (3)

ADVERSE EVENTS:
Time Frame: The adverse events were collected from October 13, 2014 thru May 16th 2017 (2 years 7 months)
Arm/Group | Luminate 1.0mg Group | Luminate 2.0mg Group | Luminate 3.0mg Group | Avastin® Group | Avastin Then Luminate 1.0 mg IVT + Sham Injection | Avastin Then Luminate 0.5 mg IVT + Sham Injection | Sham Then Luminate 1.0 mg + Avastin 1.25 mg IVT | Sham Then Luminate 0.5 mg IVT + Avastin 1.25 mg IVT | Avastin 1.25 mg + Sham IVT
All-Cause Mortality (participants affected / at risk) | 1/39 | 0/33 | 1/42 | 1/24 | 0/19 | 0/17 | 0/13 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 8/39 | 3/33 | 6/42 | 3/24 | 2/19 | 1/17 | 1/13 | 2/16 | 3/15
Other Adverse Events (participants affected / at risk) | 28/39 | 20/33 | 25/42 | 16/24 | 10/19 | 5/17 | 6/13 | 7/16 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Luminate 1.0mg Group (N=39) | Luminate 2.0mg Group (N=33) | Luminate 3.0mg Group (N=42) | Avastin® Group (N=24) | Avastin Then Luminate 1.0 mg IVT + Sham Injection (N=19) | Avastin Then Luminate 0.5 mg IVT + Sham Injection (N=17) | Sham Then Luminate 1.0 mg + Avastin 1.25 mg IVT (N=13) | Sham Then Luminate 0.5 mg IVT + Avastin 1.25 mg IVT (N=16) | Avastin 1.25 mg + Sham IVT (N=15)
Infections and infestations (Infections and infestations) | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2
Cardiac disorders (Cardiac disorders) | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0
eye disorders (Eye disorders) | 3 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Metabolism and nutritional disorders (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasms benign malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nervous system disorder (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Renal and urinary disorders (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respitatory, thoracic and mediastinal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Surgical and medical procedures (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
general disorders (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vascular disorders (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luminate 1.0mg Group (N=39) | Luminate 2.0mg Group (N=33) | Luminate 3.0mg Group (N=42) | Avastin® Group (N=24) | Avastin Then Luminate 1.0 mg IVT + Sham Injection (N=19) | Avastin Then Luminate 0.5 mg IVT + Sham Injection (N=17) | Sham Then Luminate 1.0 mg + Avastin 1.25 mg IVT (N=13) | Sham Then Luminate 0.5 mg IVT + Avastin 1.25 mg IVT (N=16) | Avastin 1.25 mg + Sham IVT (N=15)
Blood and Lymphatic (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders (Cardiac disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
eye disorders (Eye disorders) | 17 (18) | 9 (9) | 11 (20) | 7 (19) | 6 (7) | 1 (1) | 4 (9) | 5 (6) | 1 (1)
gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
infections and infestations (Infections and infestations) | 6 (6) | 5 (5) | 4 (5) | 3 (3) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 5 (5) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations (Investigations) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutritional disorders (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (5) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
musculoskeletal and connective tissue (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
psychiatric disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders (Vascular disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator will submit to Sponsor a copy of the proposed publication or presentation and the name of the scientific journal or forum to which it will be submitted- at least ninety (90) days prior to the submission.Investigator shall comply with Sponsor's request to delete references to Confidential Information,in any such paper or presentation and agrees to withhold publication or presentation of same for an additional ninety (90) days in order to permit Sponsor to obtain patent protection.

DOCUMENTS (2):
  • Study Protocol (2016-03-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT02348918/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT02348918/SAP_001.pdf